CLINICAL TRIAL: NCT06177561
Title: Safety and Efficacy of LPE in Clearing DSA in Patients Who Received Allo-HSCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RuijinLjm1
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-11

CONDITIONS: Leukemia
Keywords: lymphoplasma exchange,LPE; donor specific antibody,DSA; allogeneic hematopoietic stem cell transplantation，allo-HSCT; graft failure,GF; graft-versus-host disease，GVFHD
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LPE group (Experimental): 1. Serum DSA positive: MFI ≥ 2000；Between the ages of 18 and 65, male and female are not limited；Planned to undergo allo-HSCT , with an estimated survival time of>3 months and an ECOG physical fitness score of 0-2；Normal renal function (BUN, Cr ≤ 1.5 times the upper limit of normal value, Ccr>80ml/min)
  2. Normal liver function (defined as ALT and AST ≤ 1.5 times the upper limit of normal
  3. TBiL ≤ 1.5 times the upper limit of normal)
  4. ECG did not indicate any AMI, arrhythmia, or IAVB
  5. No CI (defined as LVEF ≥ 50%, normal MYO and BNP)
  6. Non active RHD
  7. Chest X-ray or physical examination did not indicate cardiac dilatation
  8. Normal lung function (defined as FEV1, FVC, DLCO ≥ 60% predicted value).
  Interventions: Procedure: Lymphoplasma exchange

INTERVENTIONS:
Procedure: Lymphoplasma exchange — The LPE treatment regimen is: LPE*2 times (20-30ml/kg, treatment interval of 2 days);CD20 monoclonal antibody 375mg/m2*2 times, gamma globulin 0.4g/kg/d*5d.

SUMMARY:
The aim of this study is to prospectively explore the effectiveness and safety of LPE in clearing DSA, and to investigate the clinical efficacy of a combination therapy with LPE in patients undergoing genetic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
We recruited 38 patients according to the inclusion criteria.(Inclusion criteria: 1. Serum DSA positive: MFI ≥ 2000；Between the ages of 18 and 65, male and female are not limited；Planned to undergo allo-HSCT , with an estimated survival time of>3 months and an ECOG physical fitness score of 0-2；Normal renal function (BUN, Cr ≤ 1.5 times the upper limit of normal value, Ccr>80ml/min). 2. Normal liver function (defined as ALT and AST ≤ 1.5 times the upper limit of normal. 3. TBiL ≤ 1.5 times the upper limit of normal). 4. ECG did not indicate any AMI, arrhythmia, or IAVB. 5. No CI (defined as LVEF ≥ 50%, normal MYO and BNP). 6. Non active RHD. 7. Chest X-ray or physical examination did not indicate cardiac dilatation. 8. Normal lung function (defined as FEV1, FVC, DLCO ≥ 60% predicted value).)

Sample the peripheral blood of the patient at four timepoints（Before LPE treatment (D0); Before stem cell transfusion; On the 10th day of stem cell transfusion;On the 30th day of stem cell transfusion).Using multiplex bead analysis on the Luminex platform (Luminex Corporation, Austin, TX, USA), including the LAB screening PRA and LAB screening hybrid method, all patients' ethylenediamine tetraacetic acid (EDTA)-treated serum was tested for anti-HLA class I and class II antibodies.According to the manufacturer's instructions, the semi-quantitative measurement of DSA levels was performed by LAB screening single antigen beads assay (One Lambda; ThermoFisher), and the results were expressed as MFI.The cumulative DSA MFI was calculated by summing the MFI of all detected DSA under HLA antigen resolution.

Evaluate the effectiveness of LPE by comparing it with the historical control group that has undergone TPE treatment in the past

ELIGIBILITY:
Inclusion Criteria:

1. Serum DSA positive: MFI ≥ 2000；Between the ages of 18 and 65, male and female are not limited；Planned to undergo allo-HSCT , with an estimated survival time of>3 months and an ECOG physical fitness score of 0-2；Normal renal function (BUN, Cr ≤ 1.5 times the upper limit of normal value, Ccr>80ml/min)
2. Normal liver function (defined as ALT and AST ≤ 1.5 times the upper limit of normal
3. TBiL ≤ 1.5 times the upper limit of normal)
4. ECG did not indicate any AMI, arrhythmia, or IAVB
5. No CI (defined as LVEF ≥ 50%, normal MYO and BNP)
6. Non active RHD
7. Chest X-ray or physical examination did not indicate cardiac dilatation
8. Normal lung function (defined as FEV1, FVC, DLCO ≥ 60% predicted value)

Exclusion criteria：

1. Patients with severe allergies to blood products
2. The following comorbidities exist: active infection patients, active rheumatism patients
3. Patients with secondary immunoglobulin deficiency
4. Serious damage to important organ functions, such as respiratory failure, heart failure, decompensated liver dysfunction, renal dysfunction, etc
5. Unable to obtain informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-11-08 (Estimated); Study Completion 2025-11-08 (Estimated)

PRIMARY OUTCOMES:
The degree of decrease in DSA | Before LPE treatment (D0); Before stem cell transfusion; On the 10th day of stem cell transfusion；On the 30th day of stem cell transfusion
  A semiquantitative measurement of the DSA level was performed by LAB screen single antigen bead assays (One Lambda; Thermo Fisher) and the results were expressed as MFI

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxia Hu, Dr, Principal Investigator — Ruijin Hospital; Xuefeng Wang, Dr, Principal Investigator — Ruijin Hospital; Zilu Zhang, Dr, Principal Investigator — Ruijin Hospital; Xiaohong Cai, Dr, Principal Investigator — Ruijin Hospital; Xi Wu, Dr, Principal Investigator — Ruijin Hospital; Jialu Zhao, bachelor, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
We will protect the personal information of the subjects